CLINICAL TRIAL: NCT04193488
Title: Comparison of Analgesic Efficacy of Mid-Transverse Process to Pleural (MTP) Block and Erector Spinal Plan (ESP) Block in Spinal Surgery
Brief Title: Mid-Transverse Process to Pleural (MTP) Block and Erector Spinal Plan (ESP) Block in Spinal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gulhane School of Medicine (Other)
Responsible Party: Principal Investigator, Mehmet Burak Eşkin, Assistant Professor, Gulhane School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19/342
Record Dates: First submitted 2019-12-04; First posted 2019-12-10 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Postoperative Pain; Anesthesia, Regional; Spinal Stenosis
Keywords: spinal surgery; Erector spina plan block; Mid-transverse process to pleura block; post-operative analgesia
MeSH Terms: conditions — Pain, Postoperative; Spinal Stenosis

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to 30 patients with MTP block (Group MTP) and 30 patients with ESP block (Group ESP) and 30 patients with no block (Group K) in addition to patient-controlled analgesia (PCA).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MTP block (Group MTP) (Active Comparator): In the MTP Group, a high frequency HFL-50 15-6 MHz linear ultrasound probe will be placed vertically approximately 3 cm laterally from the midpoint of the incision line in the midline. Using the parasaggital scan, the block needle (50 mm 22 Gauge will be advanced from the caudal to the cervical target of the paravertebral space. When the needle tip reaches the midpoint between the transverse process and the pleura, 1 ml normal saline is performed. Once the needle tip has been confirmed, 20 ml of 0.25% bupivacaine will be given to the block. The same procedure will be applied 3 cm later than the incision line.
  Interventions: Behavioral: MTP block
- ESP block (Group ESP) (Active Comparator): In the ESP group, a high-frequency 15-6 megahertz linear ultrasound probe will be placed vertically approximately 3 cm laterally from the midpoint of the incision line in the midline. Once the erector spinae muscle and transver projections have been identified, the peripheral nerve blockage needle (50 mm 22 Gauge) will be advanced from caudal to cranial between the fascia of the erector spina muscle and the transverse process. After 1 ml normal saline injection, this plane will open. Twenty milliliters of 0.25% bupivacaine will be given for the block. The same procedure will be applied from the other 3 cm lateral of the incision line.
  Interventions: Behavioral: ESP block
- no block (Group C) (Active Comparator): No regional plan block will be applied to the control group. Conventional analgesic methods were applied.
  Interventions: Behavioral: No Block group

INTERVENTIONS:
Behavioral: MTP block — In the MTP Group, a high frequency HFL-50 15-6 MHz linear ultrasound probe will be placed vertically approximately 3 cm laterally from the midpoint of the incision line in the midline. Using the parasagital scan, the block needle (50 mm 22 Gauge) will be advanced from the caudal to the cervical target of the paravertebral space. When the needle tip reaches the midpoint between the transverse process and the pleura, 1 ml saline is performed. Once the needle tip has been confirmed, 20 ml of 0.25% bupivacaine will be given to the block. The same procedure will be applied 3 cm later than the incision line.
  Arms: MTP block (Group MTP)
Behavioral: ESP block — In the ESP group, a high-frequency 15-6 megahertz linear ultrasound probe will be placed vertically approximately 3 cm laterally from the midpoint of the incision line in the midline. Once the erector spinae muscle and transver projections have been identified, the peripheral nerve blockage needle (50 mm 22 Gauge) will be advanced from caudal to cranial between the fascia of the erector spina muscle and the transverse process. After 1 ml saline injection, this plane will open. Twenty milliliters of 0.25% bupivacaine will be given for the block. The same procedure will be applied from the other 3 cm lateral of the incision line.
  Arms: ESP block (Group ESP)
Behavioral: No Block group — No regional plan block will be applied to the control group. Conventional analgesic methods were applied.
  Arms: no block (Group C)

SUMMARY:
Ethics committee approval was taken on October 22, 2019, numbered 19/342. 120 adult patients who will undergo spine stabilization surgery between October 2019 and January 2020 in "Gülhane Training and Research Hospital" were planned to be included in the study. Patients will be randomized to 30 patients with MTP block (Group MTP) and ESP block (Group ESP) and no block (Group K) in addition to patient-controlled analgesia (PCA). Postoperative pain scores, analgesic use, number of PCA button presses, total amount of opioid administered and complications due to opioids will be recorded. The obtained data will be compared statistically.

DETAILED DESCRIPTION:
Ethics committee approval was taken on October 22, 2019, numbered 19/342. 120 adult patients who will undergo spine stabilization surgery between October 2019 and January 2020 in Gulhane Training and Research Hospital were planned to be included in the study. Appropriate patients will be informed about the study and their written consent will be obtained. All patients were scheduled for ASA I-III. Exclusion criteria for patients are as follows: ≤18 or ≥81 years old, body mass index (BMI) ≥30 or ≤18 kg / m2, skin infection where the needle is punctured, allergic drugs to any of the study, pre-existing pain syndromes, pregnancy, severe liver diseases), kidney diseases (serum creatinine greater than 2 mg / dL, oliguria, anuria or hemodialysis) or cardiovascular disorders (functional class of the New York Heart Association greater than III). During the preoperative visit, all patients will be instructed on how to assess their pain using a numerical analogue pain scale (0 = no pain, 10 = maximum pain to be considered) and patient-controlled analgesia (PCA). Patients will be randomized according to a computer-generated random number table, in addition to patient-controlled analgesia (PCA) with MTP block (Group MTP) and ESP block (Group ESP) and no block (Group K). Nerve blocks will be made at the end of the operation after the surgical site is sutured and intact before the dressing is done. The linear ultrasound probe will be applied in the prone position bilaterally in the region of the transverse process corresponding to the center of the incision line by the same three experienced senior doctors with ultrasound guidance covered with sterile probe sheath. In the ESPB group, a high-frequency 15 6 MHz (Megahertz) linear ultrasound probe will be placed vertically about 3 cm laterally from the midpoint of the incision line in the midline. Once the erector spinae muscle and transverse projections have been identified, the peripheral nerve blockage needle (50 mm 22 Gauge) will be advanced from caudal to cranial between the fascia of the erector spina muscle and the transverse process. After 1 ml normal saline injection, this plane will open. Twenty milliliters of 0.25% bupivacaine will be given for the block. The same procedure will be applied 3 cm later than the incision line. In the MTP Group, a high frequency HFL-50 15-6 MHz linear ultrasound probe will be placed vertically approximately 3 cm laterally from the midpoint of the incision line in the midline. Using the parasaggital scan, the block needle (50 mm 22 Gauge) will be advanced from the caudal to the cervical target of the paravertebral cavity. When the needle tip reaches the midpoint between the transverse process and the pleura, 1 ml normal saline is performed. Once the needle tip has been confirmed, 20 ml of 0.25% bupivacaine will be given to the block. The same procedure will be applied 3 cm later than the incision line.

No regional plan block will be applied to the control group. All groups will receive analgesia in the postoperative period using patient-controlled analgesia (PCA), and the pain will be evaluated three days postoperatively using a numerical grading scale (NRS) ranging from 0 (painless) to 10 (worst imaginable pain). The number of PCA button presses, the total amount of opioids applied, and complications associated with opioids will be recorded. The obtained data will be compared statistically

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years old
* ASA (American Society of Anesthesiologists) score between I-III.

Exclusion Criteria:

* ASA (American Society of Anesthesiologists) score >III,
* emergency surgery,
* secondary surgery,
* receiving chronic pain treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-10-23 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
numeric rating scale (NRS) | three days postoperatively
  Pain 0 (no pain) to 10 (worst pain imaginable), ranging from a numeric rating scale (NRS) was assessed using three days after surgery
use of patient control analgesia | three days postoperatively
  The number of PCA button presses, the total amount of opioids applied
complications related to opioids | three days postoperatively
  Nausea, Vomiting, Itching, Constipation, Difficulty in urination, Difficulty in Concentration, Drowsiness or difficulty staying awake, Feeling of light dizziness, Feeling of dizziness, Feelings of general fatigue or weakness, Dry mouth, Headache
Additional analgesic use | three days postoperatively
  Additional analgesic dexketoprofen (trometamol) 50 mg / 2 ml will be administered to patients with an NRS score> 3 and the amount of use will be recorded.analgesics

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet B EŞKİN, Study Director — Gulhane Training and Research Hospital; Ayşegül Ceylan, Principal Investigator — Gulhane Training and Research Hospital
Locations (1):
- Gulhane Training and Research Hospital, Ankara, Keçiören, Turkey (Türkiye)